CLINICAL TRIAL: NCT04871126
Title: Predictive Value of Inflammatory Indexes and CHA2DS2-VASc Score for Left Ventricular Thrombus in Acute Anterior Myocardial Infarction With Left Ventricular Dysfunction
Brief Title: Predictive Value of Inflammatory Indexes and CHA2DS2-VASc Score for LVT in ANT-MI With Left Ventricular Dysfunction
Status: Completed | Type: Observational
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHA2DS2-VASc score
Record Dates: First submitted 2021-04-25; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Left Ventricular Thrombus; Acute Anterior Myocardial Infarction; Left Ventricular Dysfunction
Keywords: left ventricular thrombus;anterior myocardial infarction; Risk factors
MeSH Terms: conditions — Anterior Wall Myocardial Infarction; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LVT group: left ventricular thrombus in acute anterior myocardial infarction patients with left ventricular dysfunction
  Interventions: Other: inflammatory indexes and CHA2DS2-VASc score
- non-LVTgroup: acute anterior myocardial infarction patients with left ventricular dysfunction while without LVT
  Interventions: Other: inflammatory indexes and CHA2DS2-VASc score

INTERVENTIONS:
Other: inflammatory indexes and CHA2DS2-VASc score — inflammatory indexes and CHA2DS2-VASc score

SUMMARY:
To investigate the predictive value of inflammatory indexes and CHA2DS2-VASc score for anterior myocardial infarction (ANT-MI) with left ventricular thrombus(LVT) (LVT).

DETAILED DESCRIPTION:
The clinical data were collected from 371consecutive patients with ANT-MI in our hospital from January 2014 to January 2021.As a result,totally 62 patients with LVT were selected as the experimental group and 186 patients with non-LVT as the control group .The observation indexes included baseline data, coronary angiography, disease course, laboratory examination and auxiliary examination.Patients with severe organic disease and having previous history of left ventricular aneurysm( LVA) and LVT were excluded.Data was analyzed by software SPSS 22.0 for statistical analysis,and the logistic regression model was established.A P<0.05 was considered statistically significant, and the risk factors of LVT formation were retrospectively analyzed.

ELIGIBILITY:
Inclusion Criteria:

acute anterior myocardial infarction with left ventricular dysfunction

Exclusion Criteria:

end-stage organic disease, thrombotic hematological disorders, previous anticoagulant use, and poor echogenicity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included a total of 371 patients with anterior myocardial infarction (ANT-MI) treated with emergency prior percutaneous coronary intervention (pPCI) in our hospital betweenfrom January 2014 andto January 2021. Patients were eligible for enrollmentenrolment if they had a reduced left ventricularLV ejection fraction (LVEF) ( ≤40%). and if detailed data on demographic and clinical characteristics were documented. Exclusion criteria were end-stage organic disease, thrombotic hematological disorders, previous anticoagulant use, and poor echogenicity (Figure 1). Based on the study criteria, 123 patients were excluded from the study; thus, 248 patients were included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
the predictive of the inflammatory indexes and CHA2DS2-VASc score in LVT | Day 1
  the logistic regression model was established between the indexes and LVT

IPD SHARING:
Plan to Share IPD: Undecided